CLINICAL TRIAL: NCT05034081
Title: Impact Of Post-Bariatric Body Contouring Procedures on Patient Body Weight and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Shadad Rateb Mohamed, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AUN
Record Dates: First submitted 2021-08-18; First posted 2021-09-05 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric; Weight regain; Metabolism
MeSH Terms: interventions — Body Contouring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): to know the effect of post-bariatric body contouring surgery on weight loss and metabolism
  Interventions: Procedure: body contouring
- group B (No Intervention): compare this group of patients with group A to detect weight changes and metabolic changes without any post-bariatric intervention

INTERVENTIONS:
Procedure: body contouring — any post-bariatric body contouring surgery included
  Arms: group A

SUMMARY:
Is post-bariatric body contouring surgery prevent weight regain or no, and what is the effect on the patient's Metabolism? Few literature studies report body contouring surgery to be positively associated with maintained weight loss after obesity surgery but the measures of outcomes are diverse, and the collective magnitude of such an association is unknown.

The changes in gastrointestinal hormones, adipokines, and cytokines as well as in hypothalamic neuropeptides and neurotransmitters resemble the changes observed in the anorexia/cachexia, suggesting that bariatric surgery triggers a catabolic state responsible for loss of appetite and prolonged body weight reduction.

Weight regain after gastric bypass surgery occurs in about half of all patients within 2 years. About 50% of patients eventually gain a little weight back after hitting their low point. We need a more thorough evaluation to determine what factors - medical, psychological, lifestyle - are involved in the weight gain. One of the factors that seem to be responsible for the degree and durability of weight loss is post-bariatric body contouring procedures. However, metabolic consequences of removing excess subcutaneous adipose tissue by body contouring procedures have to a lesser extent been explored

ELIGIBILITY:
Inclusion Criteria:

* Post-bariatric (sleeve) patients will do body contouring surgery.
* Post-bariatric patients has been stable within 5 kg for 3 months
* Age between 20-60 years old.
* patients use the determinant fixed diet.

Exclusion Criteria:

* Age below 20 and above 60 years old.
* Non-compliance with the fixed diet.
* psychotic patients.
* Female patients seeking pregnancy.
* Endocrine causes of obesity.
* Bariatric surgery other than sleeve.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
weight changes by kilograms | 4 years
  to know the effect of post-bariatric body contouring surgery in weight. Detect the weight cahnges of the patient every month afer body contouring surgery and body mass index also measured every month for six months
Level of Tumor necrotizing factor alfa in blood | 4 years
  Its a clinical laboratory investigation will be done before the body contouring surgeries and 3 and 6 months after. Tumor necrotizing factor alfa increase afer bariatric surgery and we want to know if its complete on increasing after body contouring surgeries or decresae . Tnf-a is measured by pg/ml
Level of BNP in blood | 4 years
  Its a clinical laboratory investigation will be done before the body contouring surgeries and 3 and 6 months after. BNP highly increase with catabolism after bariatric surgery and we want to know the effect of body contouring surgeries in the level of BNP. BNP unit is pg/ml
Level of high sensitive CRP in blood | 4 years
  Its a clinical laboratory investigation will be done before the body contouring surgeries and 3 and 6 months after. hsCRP increase with catabolism after bariatric surgery and we want to know the effect of body contouring surgeries in blood level of hsCRp. The unit of hsCRP is mg/dl.

SECONDARY OUTCOMES:
Patient satisfaction score | 4 years
  From 1 to 5 .
  1 very dissatisfied 5 very satisfied Increase in number means increase satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shadad, Master, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
It will be shared as numbers and the name of participants will not shared